CLINICAL TRIAL: NCT00826293
Title: The Clinical Efficacy of Belting Stabilization for Shoulder Pain: A Double Blinded Randomized Clinical Trial
Brief Title: The Clinical Efficacy of Belting Stabilization for Shoulder Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Helen Razmjou, Dr. Helen Razmjou, Physical Therapist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 224-2008
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Rotator Cuff Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- True Stabilization Group (Active Comparator): Patients will be randomized to one of the two treatment groups (true stabilization vs. sham stabilization). Patients will be exercising with a belt that is expected to reduce impingement of the rotator cuff tendons.
  Interventions: Procedure: Stabilization belt
- Sham Stabilization (Sham Comparator): Patients receive sham stabilization. The sham procedure imitates the treatment without any true effect.
  Interventions: Procedure: Stabilization belt

INTERVENTIONS:
Procedure: Stabilization belt — Patients receive true stabilization.
  Other Names: Belt Stabilization
  Arms: True Stabilization Group
Procedure: Stabilization belt — Patients receive sham stabilization.
  Other Names: Ineffective stabilization
  Arms: Sham Stabilization

SUMMARY:
Application of a belt for stabilization while exercising accelerate and optimize recovery in patients diagnosed with shoulder impingement syndrome.

DETAILED DESCRIPTION:
Stabilization through belts is commonly used as an adjunct for treatment of musculoskeletal problems. Although this treatment is popular among clinicians, there is a paucity of evidence on its use for shoulder pathology. The objective of this double-blinded longitudinal randomized controlled trial (RCT) is to determine the clinical efficacy of stabilization belting applied to patients receiving rehabilitation treatment for shoulder impingement syndrome. The study population will include patients who have been referred to the physiotherapy department of the Holland Orthopaedic & Arthritic Centre for conservative treatment. Patients will be randomized into the treatment and control groups. The primary outcome measure is the Quick Disabilities of Arm, Shoulder and Hand (QuickDASH) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of impingement syndrome or post-surgical stiffness with an abnormal scapulothoracic rhythm

Exclusion Criteria:

* Inability to speak or read English
* Evidence of major joint trauma causing fracture
* Infection
* Underlying metabolic or inflammatory disease
* Avascular necrosis
* Frozen shoulder
* Major medical illness
* Psychiatric illness that precluded informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-01; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The Primary outcome measure is a subjective measure, the Quick Disability of the Arm, Shoulder and Hand (QuickDASH) | Outcome measures are collected before the initial treatment, at 3 weeks, and at 6 weeks following the initial treatment

SECONDARY OUTCOMES:
The secondary subjective outcomes include a joint specific measure, the American shoulder and Elbow Surgeons (ASES) score, and the work limitation questionnaire (WLQ-25). | Outcome measures are collected before the initial treatment, at 3 weeks, and at 6 weeks following the initial treatment

CONTACTS AND LOCATIONS:
Overall Officials: Helen Razmjou, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Holland Orthopaedic and Arthritic Centre, Toronto, Ontario, Canada